CLINICAL TRIAL: NCT06860256
Title: Comparison of the Effects of Different Exercise Training Programs on Dysmenorrhea Symptoms, Sleep and Quality of Life in University Students with Primary Dysmenorrhea
Brief Title: Different Exercise Training Programs in University Students with Primary Dysmenorrhea
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Gizem Tas Gecit, PhD student, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HasanKU-FTR-GTG-01
Record Dates: First submitted 2025-02-14; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Exercise; Primary Dysmenorrhea
Keywords: primary dysmenorrhea; exercises
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Exercise intervention in three groups
Who Masked: Participant
Masking Description: We aim to present the effects of Basic Body Awareness Therapy, High Intensity Interval Training and Classical exercise training and lifestyle recommendations on parameters such as dysmenorrhea symptoms, sleep and quality of life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Basic Body Awareness Therapy (Active Comparator): Basic Body Awareness Therapy (TBFT) is a physiotherapy modality that focuses on improving the health and well-being of patients with mental health problems and/or psychosomatic and chronic pain, long-term musculoskeletal and neurological disorders. In TBFT sessions, physiotherapists improve the patient's contact with "self" by focusing on basic movement principles while performing simple daily movements such as lying, sitting, standing, walking, use of sound and massage. Mental awareness, postural balance and free breathing are considered key elements. The pparticipants is invited to explore and integrate flow, rhythm and intentionality in coordinated movements in relation to time, space and energy. TBFT is practiced 2 days a week, 60 minutes, 5-12 weeks, depending on the patient.
  Interventions: Other: Basic Body Awareness Therapy
- High Intensity Interval Training (HIIT) (Active Comparator): High Intensity Interval Training (HIT) is a protocol filled with exercises that challenge the body and increase the heart rate, unlike normal cardio methods. The most commonly used of these protocols is the Tabata protocol. The Tabata protocol involves the re-synthesis of ATP through anaerobic and aerobic processes during high intensity exercises lasting more than a few seconds. Tabata can be done on a running track, in nature, in water, in a gym or with training aids such as stationary bicycles, jump ropes, sandbags, etc. HWCA improves metabolic functions and cardiovascular system. Recent studies have shown that High intensity interval training improves adaptation, health and performance parameters in athletes and individuals with a normal lifestyle (sedentary).Tabata exercise protocol is an 8 repetition training program with 20 seconds of work and 10 seconds of rest. Warm-up and cool-down exercises of 5 minutes each should be performed to prevent injuries and negativities.
  Interventions: Other: High Intensity Interval Training
- Classical Exercise (CE) and Lifestyle Recommendations (LSS) (Active Comparator): Classical Exercise (CE) and Lifestyle Recommendations (LSS), classical exercises used in PD include abdominal, pelvic floor muscles, hip flexors, and whole body stretches (13).Non-pharmaceutical strategies for pain management in LSS include adopting relaxation (rest, warm-up, massage, music, etc.), antalgic positions, and distraction techniques. Common techniques that facilitate relaxation and thus reduce pain include physical rest, various heat applications such as hot showers, thermal seed packs, electric blankets, and drinking warm herbal teas such as chamomile tea.
  Interventions: Other: Classic Exercise and Lifestyle Tips

INTERVENTIONS:
Other: Basic Body Awareness Therapy — In TBFT sessions, physiotherapists improve the patient's contact with "self" by focusing on basic movement principles while performing simple daily movements such as lying, sitting, standing, walking, use of sound and massage. Mental awareness, postural balance and free breathing are considered key elements. The patient is invited to explore and integrate flow, rhythm and intentionality in coordinated movements in relation to time, space and energy. TBFT is practiced 2 days a week, 60 minutes, 5-12 weeks, depending on the patient.
  Arms: Basic Body Awareness Therapy
Other: High Intensity Interval Training — Tabata exercise protocol is an 8 repetition training program with 20 seconds of work and 10 seconds of rest. Warm-up and cool-down exercises of 5 minutes each should be done to prevent injuries and negativities. Although the application varies according to the patient, YŞİA is applied 2 days a week, 15-30 minutes, in processes ranging between 2-12 weeks.
  Arms: High Intensity Interval Training (HIIT)
Other: Classic Exercise and Lifestyle Tips — Classical Exercise (CE) and Lifestyle Recommendations (LSR), Classical exercises used in PD include abdominal, pelvic floor muscles, hip flexors, whole body stretching. Non-pharmaceutical strategies for pain management in LRS include adopting relaxation (rest, warm-up, massage, music, etc.), antalgic positions, and distraction techniques. Common techniques that facilitate relaxation and thus reduce pain include physical rest, hot showers, various heat applications such as thermal seed bags, electric blankets, and drinking hot herbal teas such as chamomile tea.
  Arms: Classical Exercise (CE) and Lifestyle Recommendations (LSS)

SUMMARY:
Dysmenorrhea is severe lower abdominal pain in women during menstruation. The pain is usually cramping and can radiate to the thighs or lower spine. Lower abdominal pain may be accompanied by vomiting, headache, back pain, diarrhea, fatigue, etc. Depending on the pathophysiology, dysmenorrhea is classified into two types: primary and secondary. Primary dysmenorrhea (PD) is menstrual pain associated with normal ovulatory cycles in the absence of pelvic pathology and a clear physiologic etiology and is most commonly seen in adolescents and young adults. There are numerous studies on PD in the literature, but there is still a lack of studies on which of the non-pharmacologically recommended exercise and other methods is more effective on dysmenorrhea symptoms, sleep and quality of life for individuals with this problem. Different exercise intensities may affect PD symptoms through different mechanisms. Moderate to high intensity exercise may reduce pain by increasing anti-inflammatory cytokines, whereas less intense exercise, such as yoga, affects pain levels by decreasing cortisol levels. The lack of research on which exercise training is more effective in PD individuals was considered as a limitation. In the light of this information, the aim of the investigators study is to compare the effects of different training techniques on dysmenorrhea symptoms, sleep and quality of life in PD treatment and to present the preferability of these techniques based on evidence.

DETAILED DESCRIPTION:
Dysmenorrhea is severe lower abdominal pain in women during menstruation. The pain is usually cramping and can radiate to the thighs or lower spine. Lower abdominal pain may be accompanied by vomiting, headache, back pain, diarrhea, fatigue, etc. Depending on the pathophysiology, dysmenorrhea is classified into two types: primary and secondary. Primary dysmenorrhea (PD) is menstrual pain associated with normal ovulatory cycles in the absence of pelvic pathology and a clear physiologic etiology and is most common in adolescents and young adults. Secondary dysmenorrhea is menstrual pain associated with an identifiable disease (endometriosis, fibroids, adenomyosis, pelvic adhesions, polyps in the endometrium, pelvic inflammatory disease) or intrauterine contraceptive use. PD usually occurs only one or two years after menarche. Menstrual pain starts a few hours before or during menstruation and lasts for 2-3 days. The pain is most severe in the first 24-36 hours of menstruation.

According to the World Health Organization, 94% of girls aged 10-20 and 8.8% of women aged 19-41 suffer from menstrual cramps.It has been observed that dysmenorrhea can significantly reduce quality of life and cause absenteeism from school and work. There are different approaches to the treatment of PD. Pharmacologically, treatment is achieved through hormonal medications such as prostoglandin inhibitors, non-steroidal anti-inflammatory drugs (NSAIDs), prostoglandin inhibitors and birth control pills. Non-pharmacologically, alternative conservative treatment methods such as acupuncture and acupressure, biofeedback, heat therapies, transcutaneous electrical nerve stimulation (TENS), exercises and relaxation techniques are used because they are safe and easy to implement. PD exercise protocols include relaxation, strengthening, stretching, aerobic exercises, pelvic floor muscle strengthening exercises, yoga and pilates. Studies have shown that long-term aerobic exercises, stretching exercises and yoga relieve the symptoms of dysmenorrhea and reduce the severity of pain, but it is not known which treatment option is more effective.The investigators study will be planned as a randomized controlled trial. PD is a disease group with a high incidence especially in the 18-25 age group. Hormonal pharmacologic treatments are generally used in these patients. Although these treatments reduce symptoms, they may lead to serious contraindications in the future. In the investigators study, we aim to present the effects of Basic Body Awareness Therapy, High Intensity Interval Training, Classical exercise training and lifestyle recommendations on parameters such as dysmenorrhea symptoms, sleep and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous female university students aged 18-25 years who volunteered to participate in the study, met the criteria specified in the PD Consensus Guidelines and were diagnosed with PD by a gynecologist
* Individuals with a body mass index (BMI) between 18-35
* Individuals with a regular menstrual cycle (28 ± 7 days)
* Individuals with menstrual pain Visual Analog Scale (VAS) score of 4 cm or higher for the last 6 months

Exclusion Criteria:

* Gastrointestinal, urogynecologic, autoimmune, psychiatric, neurological diseases or other chronic pain syndromes
* Having given birth and/or being pregnant
* Intrauterine device users
* Pelvic surgery patients
* Taking oral contraceptives or medication, including antidepressants, for at least 6 months before the study
* Those with a pathological history or ultrasonography result indicating secondary dysmenorrhea
* Those who use alternative treatment methods and exercise regularly
* Serious traumatic life events that occurred in the three months prior to the start of the study
* Communication problems that may interfere with the implementation of assessments and/or treatment program

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Sociodemographic information | Two months
  Sociodemographic information, physical and other medical information about the individuals' age, weight and height will be combined to report BMI in kg/m^2 and general information about menstrual symptoms and cycles were recorded.
Menstrual Symptom Scale | Two months
  The scale consists of 22 items and is five-point Likert type. Items 1-13 belong to "Negative effects/somatic complaints" subdimension, items 14-19 belong to "Menstrual pain symptoms" sub-dimension and items 20-22 belong to "Coping methods" subdimension. The Menstrual Symptom Scale score is calculated by averaging the total score of the items in the scale. Participants are asked to assign a number between 1 (never) and 5 (always) to the symptoms they experience related to menstruation. An increase in the mean score indicates an increase in the severity of menstrual symptoms. The scale has three subdimensions. The score obtained from the subscales is calculated by averaging the total score of the items in the subscales. An increase in the mean score for the sub-dimensions indicates an increase in the severity of menstruation.
The Menstrual Attitude Questionnaire | Two months
  The Menstrual Attitude Questionnaire, is in Likert format and is rated on a scale from 1 to 7. The reliability coefficient of the original scale ranges from 0.95 to 0.97. In the Menstrual Attitude Questionnaire, higher average scores from the items, subgroups, or the overall scale indicate a "positive" attitude towards menstruation.
Evaluation of Quality of Life Short Form-12 | Two months
  Evaluation of Quality of Life Short Form-12: This questionnaire was used to evaluate quality of life, which includes 12 questions about eight domains: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health. Scoring uses the RAND system from zero to 100. The score of each domain is obtained by aggregating the question scores in every domain and dividing the resulting number by the number of questions in the same domain. A higher score indicates better quality of life.The validity and reliability of the questionnaire are approved

SECONDARY OUTCOMES:
Information About Menstruation | Two months
  To determine characteristics related to menstruation,if use of medication during menstruation, including the name, dose, amount, and timing of the medication. Additionally, individuals were assessed for the presence and severity of systemic symptoms related to menstruation.The severity of these symptoms was rated as follows: 0: None, 1: Mild, 2: Moderate, 3: Severe. This evaluation was conducted on the first day of the 1st, 2nd, and 3rd menstruation cycles.
Short-form McGill Pain Questionnaire | Two months
  A short form of the McGill Pain Questionnaire (SF-MPQ) has been developed. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Pittsburgh Sleep Quality Index | Two months
  The PSQI evaluates sleep quality and disturbances over a one-month period and consists of seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The score of each component ranges 0-3 and the global score is the sum of scores for these seven components with a range of 0-21. The global score of more than 5 indicates poor sleep quality. Developers have suggested that a global PSQI score > 5 yields a diagnostic sensitivity of 89.6% and a specificity of 86.5% in distinguishing patients with sleep problems from healthy controls in their validation study.
Epworth Sleepiness Scale | Two months
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'. The questionnaire takes no more than 2 or 3 minutes to answer.
The Stroop Test Çapa Form | Two months
  The Stroop Test is commonly used to evaluate executive functions such as selective attention and resistance to interference. The Stroop Test Çapa Form consists of three sub-sections: Stroop A, Stroop B, and Stroop C. The test involves two stimulus cards.On the first card, there are boxes in red, green, and blue colors. In the Stroop A section, the individual is asked to name the colors of the boxes as quickly as possible, following a left-to-right sequence.The second stimulus card contains the words "red," "green," and "blue" written in red, green, and blue ink colors, but the ink color and the word meaning are mismatched (e.g., the word "red" written in blue ink, the word "green" written in red ink).In the Stroop B section, the individual is asked to read the color names on this second card as quickly as possible.In the Stroop C section, instead of reading the words, the individual is instructed to name the ink color of the words as quickly as possible. During this task, the individu
State - Trait Anxiety Inventory-STAI | Two months
  The STAI state scale isscored on four levels of anxiety intensity from1 ¼ 'not at all' to 4 ¼ 'very much' and with a sumscore between 20 and 80. It is usually administeredas a self-completion questionnaire. The 20 items aredivided into two groups: ten items are formed torecord the presence of anxiety symptoms and theother ten items are scored to record the absence ofanxiety symptoms.
Heart Rate Varıabılıty Measurement To Assess Stress Level Wıth Apple Watch | Two months
  For Apple Watch users 18 and older, HRV is automatically recorded with Apple Watch (in most countries). However, you need to head to the Health app on iPhone to look at the data.Open the Health app on iPhone, tap the Browse tab in the bottom right corner, now choose Heart > Heart Rate Variability,At the top, you can change the HRV data view by day. HRV is measured manually with the Apple Watch while resting and always at the same time.
Perceived Stress Scale-10 | Two months
  The ASQ-10 scale a total of 10 items, the PSS-10 was created to measure the level of stress perceived by the individual in situations encountered in life. On a five-point Likert-type scale, participants rate each item from "Never (0)" to "Very often (4)". Items with positive statements (items 4,5,7,8) are reverse scored. A high score on the ASQ-10 scale, whose total score ranges between 0 and 40, indicates that the person's stress perception is high. The ASQ-10 scale was adapted into Turkish by Eskin et al.
Academic Stress Scale | Two months
  The 27-item scale aims to measure the general academic stress levels of university students. It consists of four sub-dimensions: difficulties in the classroom, difficulties outside the classroom, difficulties in interacting with the university and difficulties in managing different areas. The first six items of the scale belong to the difficulties in the classroom sub-dimension. The next eight items of the scale (items 7-14) belong to the difficulties outside the classroom sub-dimension. The other eight items of the scale (items 15-22) belong to the difficulties in interacting with the university sub-dimension. The last five items of the scale (items 23-27) belong to the difficulties in managing different domains sub-dimension.

CONTACTS AND LOCATIONS:
Locations (1):
- Kilis 7 Aralık University, Kilis, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I want my work to be published on international platforms.
Supporting Information: Study Protocol
Time Frame: 30 years